CLINICAL TRIAL: NCT02989987
Title: Narrative Exposure Therapy for Survivors of Sexual and Gender Based Violence in Eastern DR Congo
Brief Title: NET for SGBV Survivors in Eastern DR Congo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Vivo international e.V. (Industry)
Responsible Party: Principal Investigator, Anke Köbach, Postdoctoral Researcher, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGBV1617
Record Dates: First submitted 2016-12-06; First posted 2016-12-12 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Posttraumatic Stress Disorder; Shame
Keywords: PTSD; Shame; Narrative Exposure Therapy; Sexual and gender based violence (SGBV); DR Congo
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Coitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrative Exposure Therapy (Active Comparator): According to the NET manual (one lifeline session and 7 exposure sessions; see Schauer et al. 2011).
  Interventions: Behavioral: Narrative Exposure Therapy
- Treatment-as-usual (Active Comparator): Social support (provided on demand)
  Interventions: Behavioral: Social Support

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy
  Other Names: NET
  Arms: Narrative Exposure Therapy
Behavioral: Social Support — A local counselors provides social support on demand.
  Arms: Treatment-as-usual

SUMMARY:
Throughout the last 10 years Narrative Exposure Therapy (NET) has evolved as one of the most effective, culturally sensitive trauma interventions. In the present study the effectiveness of NET delivered by trained health personnel in a sample of survivors of sexual and gender based violence (SGBV) who suffer from Posttraumatic Stress Disorder (PTSD) will be assessed. Structured baseline, 3 and 6 month follow up interviews will be administered to assess the main outcome measures PTSD and shame. The trial will take place in Goma, DR Congo, where SGBV and its sequelae has been a major problem.

DETAILED DESCRIPTION:
Participants will be recruited through local NGOs and eligible clients randomized to the treatment (NET; app. N=100) or treatment-as-usual control (app. N=100) group, respectively. At baseline, 3-month and 6-month post-treatment, sociodemographic data, trauma exposure - esp. SGBV, PTSD, dissociation, shame, functionality and depression will be assessed in a structured interview. The interviews will be conducted by blind Congolese psychological interviewers after an intensive 3-weeks training and continuous supervision.

ELIGIBILITY:
Inclusion Criteria:

* SGBV survivors (event happened more than 4 weeks ago)
* PTSD diagnosis (DSM-5)

Exclusion Criteria:

* Acute psychosis
* Signs of cerebro-organic disease
* Acute drug or alcohol intoxication

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
PSS-I: Posttraumatic Stress Disorder symptom severity (sumscore and diagnosis) | Change from baseline to 3 and 6 months post treatment
  PTSD Symptom Scale - Interview (PSS-I; Foa & Tolin, 2000)
SVQ: Severity of shame (sumscore) | Change from baseline to 3 and 6 months post treatment
  Shame Variability Questionnaire (Brown, Rizvi & Linehan, unpublished)

SECONDARY OUTCOMES:
ShutD: Severity of Shutdown Dissociation Symptoms (sumscore) | Change from baseline to 3 and 6 months post treatment
  Shutdown Dissociation Scale (Schalinski et al., 2015)
PHQ: Depression symptom severity (sumscore) | Change in 3 and 6 months post treatment
  Patient Health Questionnaire - 9 (PHQ-9; Kroenke & Spitzer, 2002)
Functionality (sumscore) | 3 and 6 months post treatment
  Local Functionality Index (LFI; Bass et al., 2013)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Konstanz, Konstanz, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schauer, M., Schauer, M., Neuner, F., & Elbert, T. (2011). Narrative exposure therapy: A short-term treatment for traumatic stress disorders. Hogrefe Publishing.